CLINICAL TRIAL: NCT03881956
Title: The Effect of the Health-promoting Lifestyle Education Program Provided to Women With Gestational Diabetes on Maternal and Neonatal Health: A Randomized Controlled Trial
Brief Title: Health-promoting Lifestyle Education on Women With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Aslı URAL, PhD Nurse, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 443983
Record Dates: First submitted 2019-03-04; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: gestational diabetes; health-promoting lifestyle; maternal and neonatal health; education
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The study sample included 88 women (46 for the intervention and 42 for the control group) diagnosed with GDM. The control group received only usual care and they were followed according to the institution's diabetes follow-up protocol. In addition to the usual care, the intervention group was provided with an education program that consisted of three 45 min sessions.The women in the both group were administered the introductory information form, the Health-Promoting Lifestyle Profile II (HPLP-II), the Center for Epidemiologic Studies Depression Scale (CES-D) and the Short Form 36 Health Survey (SF-36) in the first assessment. After the education program, the HPLP-II, CES-D and SF-36 were re-administered to the intervention group four weeks after the first assessment. The HPLP-II, CES-D and SF-36 were re-administered to the both groups in the postpartum 6th week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with gestational diabetes (Other): 88 women with gestational diabetes (46 for the intervention group and 42 for the control group) were in the arm.
  Interventions: Behavioral: Health-promoting lifestyle education program

INTERVENTIONS:
Behavioral: Health-promoting lifestyle education program — The intervention group were included in the health-promoting lifestyle education program. The education program consisted of three 45-min sessions, which included a face-to-face lecture with the dissemination and presentation of written and visual materials. Each participant in the intervention group was given the Health-Promoting Lifestyle Booklet and the Diary of a Woman with GDM card. The booklet features all of the health-promoting practices (self-monitoring of blood glucose, nutrition, physical activity, stress, sleeping, smoking, self-care and breastfeeding). The Diary of a Woman with GDM card features the daily program that women should follow (the hours for main meals and snacks, insulin hours, etc.). The education and counseling were maintained through follow-up via phone for intervention group.

SUMMARY:
In this study the effect of the Health-Promoting Lifestyle Education Program (HPLEP) provided to women with GDM on maternal and neonatal health was investigated. The education program and also usual care applied to the intervention group, only usual care applied to the control group.

DETAILED DESCRIPTION:
The population of this study included women with GDM who received treatment in the perinatology clinic of the Istanbul Zeynep Kamil Hospital, Turkey in 2015. The records showed that 350 women with GDM were referred to the perinatology clinic in that period. The sample size was calculated using Power and Sample Size Program, with 80% power and a 0.05 margin of error, and it was determined that both the intervention and the control group should include at least 30 women with GDM. It was considered appropriate that 50 women with GDM be included in each group.

At the end of this study 46 women were in the intervention group and 42 women were in the control group.

The patients followed up in the perinatology clinic were assigned to groups through randomization (drawing lots by the clinic nurse). Data collector checked patients in the perinatology clinic daily. If there were more than one patient who met the inclusion criteria, it was determined which group to take with the lottery method. When there was only one woman with GDM in the clinic, it was determined which group to take with the lot but the next patient was taken directly to the opposite group. When two patients were in the same room, they were taken into the same group in order not to have any ethical problems. Detailed information was given to the women who met inclusion criteria and their consent was obtained using an Informed Voluntary Consent Form. The women in the both group were administered the introductory information form, the Health-Promoting Lifestyle Profile II (HPLP-II), the Center for Epidemiologic Studies Depression Scale (CES-D) and the Short Form 36 Health Survey (SF-36) in the first assessment.

The education program and also usual care applied to the intervention group. The education program consisted of three 45-min sessions, which included a face-to-face lecture with the dissemination and presentation of written and visual materials. Also each participant in the intervention group was given the Health-Promoting Lifestyle Booklet and the Diary of a Woman with GDM card. The booklet features all of the health-promoting practices (self-monitoring of blood glucose, nutrition, physical activity, stress, sleeping, smoking, self-care and breastfeeding). The Diary of a Woman with GDM card features the daily program that women should follow (the hours for main meals and snacks, insulin hours, etc.). The education and counseling were maintained through follow-up via phone for intervention group.

The women in the control group which receiving only usual care were followed according to the institution's routine diabetes follow-up protocol (monitoring blood glucose levels as frequently as indicated by the doctor, and patients are referred to dietitian and to diabetes nurse).

To assess the effectiveness of the educational program, the HPLP-II, CES-D and SF-36 were re-administered to the intervention group four weeks after the first assessment (second assessment). The HPLP-II, CES-D and SF-36 were re-administered to the both groups in the postpartum 6th week (third assessment).

ELIGIBILITY:
Inclusion Criteria:

* In gestational period of 24 to 34 weeks
* Diagnosed with GDM
* Aged 18 years or older
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of a psychiatric disease
* Multiple pregnancy
* Risk of preterm labor, placenta previa or premature rupture of the membranes
* Not volunteering to participate in the study

Ages: 19 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
Change of Health-Promoting Lifestyle Profile II (HPLP II) scores | Four weeks after randomization and within postpartum 6th week
  Primary outcome of women with GDM was their healthy lifestyle behaviours measured on the HPLP-II. This scale, developed by Walker et al. (1987) on the basis of Pender's health promotion model, measures the health-promoting behaviours associated with a health-promoting lifestyle. The scale was revised in 1996 and designated as HPLP-II (Walker et al. 1996). Bahar et al. (2008) tested the scale's validity and reliability in Turkish. The Cronbach's alpha internal consistency coefficient of the scale was found to be 0.92. Higher scores on the scale indicate a higher performance level of the determined health-promoting behaviours. The scale consists of 52 items under the six subscales of spiritual growth, nutrition, physical activity, health responsibility, interpersonal relations and stress management. The lowest and highest possible scores on the scale are 52 and 208, respectively.
Change of Short Form 36 Health Survey (SF-36) scores | Four weeks after randomization and within postpartum 6th week
  Quality of life of the women was measured using the SF-36. This scale, developed by Ware in 1987, is globally referred to as SF-36, as this acronym has been commonly used in all studies since the development of the scale. SF-36 is a self-assessment scale, consisting of 36 questions under eight subscales: physical functioning, physical role limitation, social functioning, mental health, energy-vitality, bodily pain, general health perceptions and emotional role limitation (Ware & Sherbourne 1992). Pınar (1995) tested the scale's validity and reliability in Turkish. The Cronbach's alpha internal consistency value was found to be 0.91.When the scores of each subscale in the scale increase, health-related quality of life also increases. Subscales are all separately scored. "0" point indicates poor health and "100" points states good health (Ware and Sherbourne, 1992).
Change of Center for Epidemiologic Studies Depression Scale (CES-D) scores | Four weeks after randomization and within postpartum 6th week
  CES-D Scale was used to assess symptoms of depression in women. This short scale, developed by Radloff (1977) to measure depressive symptoms, can be administered to both the general population and specially selected groups. The CES-D consists of 20 items, each of which are scored between 0 and 3. The 4th, 8th, 12th, and 16th items are reversely scored. The total score ranges between 0 and 60, and a score of 16 and higher suggests the risk of depression, while lower scores on the CES-D Scale indicate decreased risks for depression. The scale measures symptoms experienced over the most recent week of time according to frequency of occurrence, where 0= Rarely or never, 1= Sometimes, 2= Often, and 3= Usually or always. Yilmaz (2010) tested the scale's validity and reliability in Turkish. The Cronbach's alpha value was found to be 0.85 for the entire scale.
Pre-test and post-test scores | After randomization up to one week
  Women's level of knowledge about GDM was measured using pre-test and post-test question form.This form, developed by the researcher in accordance with the literature, includes questions about GDM and healthy lifestyle. There are 16 questions in the question form. The minimum score that the women in the intervention group could get from the pre-test and post-test was "0" and the maximum score was "16".

SECONDARY OUTCOMES:
Postpartum diabetes control of women | within postpartum 6th week
  Postpartum diabetes control of women with GDM was assessed through the postpartum 6th week information form that developed by the researchers on the basis of the literature.
Postpartum characteristics of neonates | in postpartum first day
  Postpartum characteristics of neonates were assessed through the neonate's information form that developed by the researchers on the basis of the literature.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03881956/Prot_SAP_000.pdf